CLINICAL TRIAL: NCT01316575
Title: Prophylactic Nasal Continuous Positive Airway Pressure (nCPAP) Following Bowel Surgery
Brief Title: Prophylactic nCPAP Following Bowel Surgery (Bio-REB File 11-27)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Royal University Hospital Foundation (Other)
Responsible Party: Principal Investigator, William McKay, Anesthesiologist, University of Saskatchewan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANES-3
Record Dates: First submitted 2011-03-07; First posted 2011-03-16 (Estimated); Results first posted 2013-02-27 (Estimated); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Postoperative Pulmonary Atelectasis; Surgery
Keywords: Continuous Positive Airway Pressure; Postoperative Complications; Respiratory Insufficiency; Colorectal Surgery
MeSH Terms: conditions — Pulmonary Atelectasis; Postoperative Complications; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nCPAP (Experimental): The experimental group will receive nasal CPAP at 10cmH20 for one hour in the Post Anesthetic Care Unit.
  Interventions: Device: nCPAP
- Low Flow Oxygen (Active Comparator): The control group will receive standard therapy of low flow oxygen via simple mask at 8 litres per minute.
  Interventions: Device: Low Flow Oxygen

INTERVENTIONS:
Device: nCPAP — The experimental group will receive nasal CPAP at 10cmH20 for one hour in the Post Anesthetic Care Unit.
  Arms: nCPAP
Device: Low Flow Oxygen — The control group will receive standard therapy of low flow oxygen via simple mask at 8 litres per minute.
  Arms: Low Flow Oxygen

SUMMARY:
The purpose of this study is to determine whether prophylactic nasal continuous positive airway pressure (nCPAP) in the post-anaesthesia care unit (PACU) improves post-operative pulmonary function following elective bowel surgery. The investigators hypothesize that one hour of nCPAP in the PACU will result in a higher partial pressure of arterial oxygen (PaO2) when compared to the standard treatment of low flow oxygen applied by face mask.

DETAILED DESCRIPTION:
Post-operative pulmonary complications, such as hypoxemia, pneumonia and respiratory failure, occur in 5-10% of patients following abdominal surgery. These post-operative pulmonary complications result in increased morbidity, mortality, ICU admission, length of hospital stay and resource use.

CPAP has shown to be an effective treatment for hypoxemia following abdominal surgery. It decreases atelectasis formation the risk of pneumonia. Application of nCPAP to treat hypoxemic respiratory failure following thoraco-abdominal surgery has shown to decrease endotracheal intubation.

Nasal CPAP has shown to be effective prophylaxis following elective cardiac and thoraco-abdominal aortic surgery. It reduces the incidence of hypoxemia, pneumonia, re-intubation and re-admission to the ICU. It has also shown to decrease the length of hospital stay.

The use of nCPAP immediately post-operatively in the PACU following abdominal surgery has not been evaluated. Nasal CPAP is better tolerated than full face mask CPAP. It allows for effective clearance of respiratory secretions, improved communication and decreases claustrophobic sensation. The PACU is a transition period from general anaesthesia into the post-operative recovery phase. During this time, residual anaesthetic causes decreased level of consciousness and sub-optimal respiratory effort. Reversal agent for neuromuscular blockade has often not reached its peak effect. Inadequate pain control may further decrease respiratory effort. This transition period may be when maximal atelectasis of alveolar lung units occurs. This time period may be optimal for the application of nCPAP for prophylaxis against hypoxemia. It may improve post-operative pulmonary function which could decrease post-operative morbidity, mortality, length of hospital stay and resource use.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo elective laparotomy for bowel surgery

Exclusion Criteria:

* age < 18 years
* postoperative admission to the intensive care unit
* a history of allergy/intolerance to Ametop

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William P McKay, MD, Principal Investigator — Professor

REFERENCES:
- [Background] Zarbock A, Mueller E, Netzer S, Gabriel A, Feindt P, Kindgen-Milles D. Prophylactic nasal continuous positive airway pressure following cardiac surgery protects from postoperative pulmonary complications: a prospective, randomized, controlled trial in 500 patients. Chest. 2009 May;135(5):1252-1259. doi: 10.1378/chest.08-1602. Epub 2008 Nov 18. PMID 19017864
- [Background] Ferreyra GP, Baussano I, Squadrone V, Richiardi L, Marchiaro G, Del Sorbo L, Mascia L, Merletti F, Ranieri VM. Continuous positive airway pressure for treatment of respiratory complications after abdominal surgery: a systematic review and meta-analysis. Ann Surg. 2008 Apr;247(4):617-26. doi: 10.1097/SLA.0b013e3181675829. PMID 18362624
- [Background] Kindgen-Milles D, Muller E, Buhl R, Bohner H, Ritter D, Sandmann W, Tarnow J. Nasal-continuous positive airway pressure reduces pulmonary morbidity and length of hospital stay following thoracoabdominal aortic surgery. Chest. 2005 Aug;128(2):821-8. doi: 10.1378/chest.128.2.821. PMID 16100174

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 4 April 2011 and ended 29 April 2012. The target enrollment was 40. 40 patients were enrolled in the study.
Period: Overall Study
Arm/Group | nCPAP | Low Flow Oxygen
Started | 20 | 20
Completed | 18 | 19
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Required alternate treatment | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | nCPAP | Low Flow Oxygen | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (12) | 61 (11.4) | 62 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 13 | 19
  Male | 14 | 7 | 21
Region of Enrollment [Number; unit: participants]
  Canada | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Alveolar - Arterial Gradient
Description: The alveolar - arterial gradient is the difference between the partial pressure of alveolar oxygen and the partial pressure of arterial oxygen
Time Frame: 1 hour following admission to PACU
Population: From the literature, a sample size of 19 subjects per group is required for a power >0.9 and alpha <0.05 assuming a normalised difference in A-a gradient between groups of 0.33 and a Standard Deviation (SD) of 0.33
Measure: Mean (Standard Deviation); unit: torr
Arm/Group | nCPAP | Low Flow Oxygen
Number analyzed (Participants) | 18 | 19
torr | 70.6 (28.3) | 134 (72.6)

2. Secondary Outcome: Number of Participants Requiring Reintubation
Time Frame: Up to 2 weeks
Measure: Number; unit: participants
Arm/Group | nCPAP | Low Flow Oxygen
Number analyzed (Participants) | 18 | 19
participants | 0 | 0

3. Secondary Outcome: Number of Participants Requiring Admission to ICU
Time Frame: Up to 2 weeks
Measure: Number; unit: participants
Arm/Group | nCPAP | Low Flow Oxygen
Number analyzed (Participants) | 18 | 19
participants | 0 | 0

4. Secondary Outcome: Length of Stay in Hospital
Time Frame: Up to 2 weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | nCPAP | Low Flow Oxygen
Number analyzed (Participants) | 18 | 19
days | 10 (7.4) | 10.9 (6.7)

ADVERSE EVENTS:
Arm/Group | nCPAP | Low Flow Oxygen
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

LIMITATIONS AND CAVEATS:
We made an assumption for FiO2, the respiratory quotient and barometric pressure in the alveolar air equation.

We did not standardize the time between extubation and application of nCPAP.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes